CLINICAL TRIAL: NCT04804683
Title: The European/International FMD Registry and Initiative (FEIRI), a Prospective Study
Brief Title: European/International FMD Registry and Initiative
Acronym: FEIRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, PERSU Alexandre, Professor, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/28AOU/464
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Fibromuscular Dysplasia
MeSH Terms: conditions — Fibromuscular Dysplasia

STUDY DESIGN:
Intervention Model Description: The study is interventional because it requires blood/urine sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort of patients with Fibromuscular Dysplasia (Other): Intervention consists in blood/urine sampling
  Interventions: Genetic: Genetic dissection of Fibromuscular Dysplasia; Other: Search for diagnostic and prognostic biomarkers of Fibromuscular Dysplasia

INTERVENTIONS:
Genetic: Genetic dissection of Fibromuscular Dysplasia — Blood sampling for genetic analysis aiming at unraveling the genetic basis of Fibromuscular Dysplasia
Other: Search for diagnostic and prognostic biomarkers of Fibromuscular Dysplasia — Blood/urine and in rare cases tissue sampling aiming at identifying biomarkers of Fibromuscular Dysplasia

SUMMARY:
The main objectives of FEIRI are:

(i) To describe the demographic and arterial characteristics of FMD and related diseases at a global scale and according to countries and/or ethnic origin

(ii) To evaluate the incidence and predictors of novel FMD lesions and complications

(iii) To explore the commonalities and differences between FMD, SCAD and so-called atypical FMD (patients with multiple dissections and/or aneurysms without string-of-beads, focal stenosis or evidence of inherited arteriopathy)

(iv) To contribute to the unravelling of genetic, proteomic and molecular mechanisms underlying FMD and related diseases

Participation to the FEIRI study implies:

(i) Collection of demographic and standard-of-care clinical data, both retrospectively (from the diagnosis of FMD to signature of the informed consent) and prospectively (on the occasion of standard-of-care follow-up).

(ii) Optional participation to a biobank implying collection of blood, urine and, in rare cases of intervention, tissue samples for genomic and proteomic analysis and identification of diagnostic and prognostic biomarkers of FMD.

Participants will be enrolled in centres from over 20 countries in Europe and beyond.

DETAILED DESCRIPTION:
Fibromuscular dysplasia (FMD) is an idiopathic, segmental, nonatherosclerotic, and noninflammatory disease of the musculature of arterial walls, leading to stenosis of small- and medium-sized arteries. FMD can be classified in multifocal FMD, characterized by alternation of stenosis and dilations ("string-of-beads") and focal FMD, corresponding to a solitary narrowing. While for long FMD was considered as a rare cause of renovascular disease mostly affecting young women, during the last decades, joint international efforts have led to a thorough reappraisal of the disease. In summary, (i) FMD is no more considered as a truly rare disease; (ii) FMD may be also diagnosed in men (10-20%) and at all ages; (iii) beyond arterial stenosis, FMD is often associated with dissections, aneurysms and arterial tortuosity; (iv) FMD is not restricted to renal arteries and often affects two or more arterial beds; (iv) multifocal FMD lesions are frequent in patients with Spontaneous Coronary Artery Dissection (SCAD).

Despite traditional views on the role of female hormones, mechanical factors and smoking, the pathophysiology of FMD remains largely unknown. In the last decade, research has been focused on genetic dissection of the disease and identification of biomarkers. Recent advances include: (i) identification of an association between FMD and an intronic variant of the Phosphatase and actin regulator 1 (PHACTR1) gene; (ii) identification of rare mutations in several genes such as Prostaglandin I2 Receptor (PTGIR) and Collagen type V alpha 1 chain (COL5A1) genes; (iii) documentation of mild Connective-Tissue Disease-like features and increased levels of Transforming Growth Factor-beta in patients with FMD; (iv) identification of a tentative proteo-genomic signature of the disease. All elements are thus in place to further dissect the pathophysiology of FMD and related diseases, refine clinical characterization, identify predictors of complications and improve screening, management and follow-up.

Unravelling the clinical characteristics, genetic and molecular basis of FMD nevertheless requires large numbers of well characterized patients. In order to address these challenges and generate new evidence pertaining to FMD and associated diseases, we aimed to create an overarching resource and study named "the European/International FMD Registry and Initiative" (acronym: FEIRI).

The objectives of FEIRI are:

To describe the demographic and arterial characteristics of FMD and related diseases at a global scale and according to countries and/or ethnic origin

To identify environmental/ hormonal factors and exposures associated with the onset and progression of FMD

To evaluate the incidence and predictors of novel FMD lesions and complications

To provide evidence-based algorithms for the diagnosis and optimal management and follow-up of patients with FMD

To explore the commonalities and differences between FMD, SCAD and so-called atypical FMD (patients with multiple dissections and/or aneurysms without string-of-beads, focal stenosis or evidence of inherited arteriopathy)

To contribute to the unravelling of genetic, proteomic and molecular mechanisms underlying FMD and related diseases

Participation to the FEIRI study implies:

Collection of demographic and standard-of-care clinical data, both retrospectively (from the diagnosis of FMD to signature of the informed consent) and prospectively (on the occasion of standard-of-care follow-up).

Optional participation (both for centres and patients) to a biobank implying collection of blood, urine and, in rare cases of intervention, tissue samples for genomic and proteomic analysis and identification of diagnostic and prognostic biomarkers of FMD.

Participants will be enrolled in centres from over 20 countries in Europe and beyond.

ELIGIBILITY:
Inclusion Criteria:

(i) Patients with established FMD, i.e at least one string-of-beads (multifocal FMD) or focal stenosis (focal FMD).

(ii) Patients with Spontaneous Coronary Artery Dissection (SCAD) in whom at least one lesion of multifocal FMD (string-of beads) in extra-coronary arteries has been identified ("SCAD-FMD").

(iii) Patients with so-called "atypical FMD" or "FMD-like presentation", i.e. patients presenting with at least one dissection or 2 aneurysms < 60-year-old, in the absence string-of-beads, focal stenosis or evidence of inherited arteriopathy.

Exclusion Criteria:

Diagnosis based only on ultrasound (need for computed tomographic angiography , magnetic resonance angiography or catheter-based angiography to confirm the diagnosis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2031-03-10 (Estimated)

PRIMARY OUTCOMES:
Wide-scale analysis of characteristics and progression of Fibromuscular Dysplasia | 10 years
  Wide-scale analysis of baseline clinical characteristics and predictors of evolution/complications of Fibromuscular Dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Persu, MD-PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No